CLINICAL TRIAL: NCT06452758
Title: Relative Energy Deficiency in Females and Males Rowers - Observational Study
Brief Title: Relative Energy Deficiency in Rowers
Status: Not yet recruiting | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: REDs2024
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Endothelial Dysfunction; Mood Disorders; Malnutrition, Calorie
Keywords: relative energy deficiency; gut permeability; rowers
MeSH Terms: conditions — Mood Disorders; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- male and female rowers: Rowers will perform 2000m ergometer test.A 2,000-m time trial is a standard test used to assess performance in rowers.
  Interventions: Other: 2000 meter ergometer test

INTERVENTIONS:
Other: 2000 meter ergometer test — Rowers will perform 2000m ergometer test. A 2,000-meter trial is a standard test used to assess performance in rowers.

SUMMARY:
This study aims to learn about relative energy deficiency in male and female rowers at the end of the direct sport preparation phase of the annual training cycle. The main questions:

- How will energy intake influence leptin, cortisol levels, mood, gut discomfort, and permeability? The observational study involves male and female rowers from the Polish rowing team.

Participants will perform 2000 meter ergometer test and 6000 ergometer test in annual training cycle. Researchers will compare outcomes from both tests.

ELIGIBILITY:
Inclusion Criteria:

* Membership in Polish Rowing Team,
* minimum five years of training,
* total training time minimum of 240 minutes,
* filling out a food diary,
* finishing 2000-meter ergometer test.

Exclusion Criteria:

* Probiotics within the last three months,
* prebiotics within the last three months
* antibiotic therapy within the last three months,
* dietary regime,
* gastrointestinal diseases.

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male rowers age 18 - 22 years.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-06-26 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
-FABP (intestinal fatty acid binding protein)to measure epithelial wall injury | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting) up to one hour after getting up, 1 minute after the test, and 3-hour recovery period
  I-FABP concentration measured in blood [ng/ml] using commercially availableenzyme-linked immunosorbent assays
Leptin to measure long-term energy balance | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting) up to one hour after getting up, 1 minute after the test, and 3-hour recovery period
  Leptin concentration measured in blood [ng/ml] using commercially availableenzyme-linked immunosorbent assays
Cortisol to measure stress | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting) up to one hour after getting up, 1 minute after the test, and 3-hour recovery period
  Stress hormone concentration measured in blood [ng/ml] using commercially available enzyme-linked immunosorbent assays
sCD14 multifunctional lipopolysaccharide receptor | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting) up to one hour after getting up, 1 minute after the test, and 3-hour recovery period
  sCD14 concentration measured in blood [ug/ml] using commercially available enzyme-linked immunosorbent assays
Claudin to measure tight junction leakage | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting) up to one hour after getting up, 1 minute after the test, and 3-hour recovery period
  Claudin concentration measured in blood [ng/ml] using commercially available enzyme-linked immunosorbent assays
POMS | day before the test
  Profile of Mood States
REST-Q sport | day before the test
  Recovery-Stress questionnaire for Athletes

SECONDARY OUTCOMES:
energy | Time Frame: whole day (24hours) before test, in the morning before the test
  energy [kcal ]of food intake measured by food diary
protein | Time Frame: whole day (24hours) before test, in the morning before the test
  protein [g ]of food intake measured by food diary
fat | Time Frame: whole day (24hours) before test, in the morning before the test
  fat [g ]of food intake measured by food diary
carbohydrate | Time Frame: whole day (24hours) before test, in the morning before the test
  carbohydrate [g ]of food intake measured by food diary
fiber | Time Frame: whole day (24hours) before test, in the morning before the test
  fiber [g ]of food intake measured by food diary
Body mass | in the morning before the test up to 1 hour after getting up
  Body mass [kg] measured by electronic scale to the nearest 0,05 kg (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan)
Body fat | in the morning before the test up to 1 hour after getting up
  Body fat [%] measured by electronic scale (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan)
Total body water | in the morning before the test up to 1 hour after getting up
  Body water [%] measured by electronic scale (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan)
Lean body mass | in the morning before the test up to 1 hour after getting up
  Lean body mass [kg] measured by electronic scale (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan)
Height | in the morning before the test up to 1 hour after getting up
  [cm] measured by high meter
Self reported scale of gastrointestinal symptoms e.g.burping, heartburn, flatulence, abdominal pain, the urge to reiterate, vomiting, diarrhoea, nausea, dizziness, and stitch | up to 1 hours after the test
  10-point scale where 10 was the symptom with the greatest severity

CONTACTS AND LOCATIONS:
Overall Officials: Anna Skarpańska-Stejnborn, Profesor, Study Director — Poznan University of Physical Education
Locations (1):
- Poznan University of Physical Education, Faculty of Sport Sciences in Gorzow, Gorzów Wielkopolski, Lubusz Voivodeship, Poland